CLINICAL TRIAL: NCT05507762
Title: A Randomized, Double-blind, Controlled Clinical Study of Human Umbilical Cord Mesenchymal Stem Cell in Patients With Cirrhosis Due to Hepatitis B (Compensation Stage)
Brief Title: Study of Human Umbilical Cord Mesenchymal Stem Cell in Patients With Cirrhosis Due to Hepatitis B (Compensation Stage)
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Renmin Hospital of Wuhan University (Other)
Collaborators: Vcanbio Cell and Gene Engineering Corp., Ltd. (Industry); Wuhan Optics Valley Zhongyuan Pharmaceutical Co., Ltd., Hubei, China (Unknown)
Responsible Party: Principal Investigator, Jiang Yingan, Principle Investigator, Clinical Professor, Renmin Hospital of Wuhan University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RenminHJiangYingan
Record Dates: First submitted 2022-08-15; First posted 2022-08-19 (Actual); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: Cirrhosis Due to Hepatitis B
Keywords: cirrhosis; compensatory stage; human umbilical cord derived mesenchymal stem cells; Cirrhosis Due to Hepatitis B
MeSH Terms: conditions — Fibrosis | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): MSCs Participants will receive antiviral drug, anti-fibrotic drugs and UC-MSCs
  Interventions: Biological: UC-MSCs
- Comparator (Placebo Comparator): Comparator participants will receive antiviral drug, anti-fibrotic drugs and saline solution
  Interventions: Biological: Saline solution

INTERVENTIONS:
Biological: UC-MSCs — Usage: The stem cell preparation in this study is used intravenously in the elbow.
  Dose: The dose of stem cell injection in this clinical study is set at 1×10^6/Kg/time per injection Duration: 5 injections per trial group for the entire duration of the course, at 1st treatment, 2-week, 4-week, 16-week, and 24-week respectively
  Arms: Experimental
Biological: Saline solution — Usage: The saline solution in this study is used intravenously in the elbow. Dose: The dose of saline solution in this clinical study is set at 250ml/time per injection Duration: 5 injections per person for the entire duration of the course, at 1st treatment, 2-week, 4-week, 16-week, and 24-week respectively
  Arms: Comparator

SUMMARY:
There are about 240 million chronic hepatitis B virus (HBV) infected people in the world, and about 2%-5% of compensated cirrhosis patients progress to decompensated cirrhosis patients every year. Studies have shown that the 5-year survival rate of decompensated cirrhosis is only 14-35%, and the quality of life and prognosis of patients are poor. Reversing or delaying the process of cirrhosis and reducing the development of compensated cirrhosis to decompensated cirrhosis is one of the effective methods for liver disease treatment. MSCs are mainly derived from bone marrow, but bone marrow mesenchymal stem cells have some shortcomings, such as cumbersome sampling, and the proliferation and differentiation ability of bone marrow mesenchymal stem cells decrease obviously with the age of donors, which is not conducive to cell therapy. Umbilical cord has many advantages, such as wide source, convenient collection, small immune rejection, and small ethical controversy, which makes it a hot spot in stem cell research and has a wider prospect in cell therapy. This clinical study will explore the efficacy and safety of human umbilical cord-derived mesenchymal stem cells in the treatment of hepatitis B virus-infected patients with compensated cirrhosis.

DETAILED DESCRIPTION:
There are about 1.7 billion people with different types of chronic liver diseases in the world, of which about 240 million are infected with chronic hepatitis B virus (HBV), and about 15%-40% of chronic hepatitis B can develop into liver cirrhosis and die of liver hardness every year There are hundreds of thousands of patients. There are about 90 million hepatitis B carriers in China, including about 20 million chronic hepatitis B carriers. Every year, about 2%-5% of compensated cirrhosis patients progress to decompensated cirrhosis patients. Studies have shown that the 5-year survival rate of decompensated liver cirrhosis is only 14-35%, and the quality of life and prognosis of patients are poor. From the progression of liver fibrosis to the decompensation of liver cirrhosis, liver failure often occurs. Statistics show that slow increase The 28-day mortality rate of patients with acute liver failure of grade 1, 2 and 3 is as high as 22%, 32% and 77%. The 90-day mortality rate was 41%, 73%, 95%. Orthotopic liver transplantation is the most effective means to treat decompensated liver failure due to liver cirrhosis, However, the shortage of donor liver, immune rejection and high cost have become treatment obstacles. Application of artificial liver support system for blood flow Plasma replacement can remove toxic substances from blood, but it can't supplement albumin and coagulation factors, and it is important to whether reducing the mortality rate is still controversial. Therefore, it reverses or delays the process of liver cirrhosis and reduces the compensatory stage of liver cirrhosis It is an important link in the treatment of liver diseases that the patients develop into decompensated stage The curative effect of medical treatment on hepatitis B cirrhosis (compensatory period) is very limited; Liver transplantation is difficult to popularize in clinical application due to the lack of donors and high cost. Mesenchymal Stem Cells (MSCs) are derived from mesoderm in early development, is a high degree of self-renewal ability, Pluripotent stem cells with high proliferation ability and multidirectional differentiation potential widely exist in bone marrow, fat, umbilical cord blood, umbilical cord, and other tissues. They can be cultured and expanded in vitro, and can differentiate into adipocytes, osteoblasts, cartilage tissues, nerve cells, hepatocytes and so on under the control of specific conditions, which has great application value in cell therapy and tissue engineering. The purpose of this study was to investigate the efficacy and safety of umbilical cord mesenchymal stem cells in the treatment of hepatitis B cirrhosis (compensatory stage). The subjects were randomly divided into two groups: umbilical cord mesenchymal stem cells injected through peripheral vein group and control group, with 10 cases in each group, a total of 20 cases. The subjects were randomly divided into two groups, namely, umbilical cord mesenchymal stem cells injected through peripheral vein group and control group. Patients in the treatment group were treated with stem cells based on conventional medical treatment. The efficacy and adverse reactions of patients were observed in detail within 24 weeks after treatment, and the long-term effect of stem cell therapy was observed after 96 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* The age is between 18 and 65 years old (including 18 and 65 years old), regardless of gender;
* The hardness of liver was detected by transient elastography, and liver cells were detected by imaging and laboratory examination There were no severe complications such as esophageal varices bleeding, ascites, or hepatic encephalopathy;
* Plasma albumin ≥ 35g / L, total bilirubin < 35μThe activity of prothrombin was more than 60%, The child Pugh score was Grade A;
* Willing to participate in this clinical study, will cooperate with doctors to carry out research, and sign informed consent.

Exclusion Criteria:

* Spontaneous peritonitis or other severe infections were found;
* Patients with hepatorenal syndrome;
* Severe hepatic encephalopathy, massive hemorrhage of digestive tract or variceal hemorrhage occurred;
* Combined with serious heart, lung, kidney, blood, endocrine system diseases; There were portal vein thrombosis;
* Patients with positive serum HIV antibody;
* The etiology of liver cirrhosis is not chronic HBV infection (HCV, EBV, CMC, autoimmune liver disease, primary biliary cirrhosis, parasitic, alcoholic, drug-related, genetic metabolic, genetic metabolic diseases), or other factors besides chronic HBV infection;
* Malignant tumor of liver or other organs;
* Pregnant women, lactating women, or those with recent birth planning;
* Those who have a history of alcoholism and drug abuse and fail to give up effectively;
* Participated in other clinical trials within 3 months before enrollment;
* Participated in stem cell clinical research before;
* Not willing to sign informed consent form;
* Those who have neurological or mental disorders and are unable to cooperate or are unwilling to cooperate;
* Other situations in which the researcher considered that the patient should not participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-07-20 (Actual); Primary Completion 2023-07-20 (Estimated); Study Completion 2023-08-20 (Estimated)

PRIMARY OUTCOMES:
FibroScan | Change from Baseline Liver stiffness at week 24
  Parameters of liver stiffness
IV-C | Change from Baseline at week 24
  Change of Serum hepatic fibrosis indexes
HA | Change from Baseline at week 24
  Change of Serum hepatic fibrosis indexes
LN | Change from Baseline at week 24
  Change of Serum hepatic fibrosis indexes
PC-III | Change from Baseline at week 24
  Change of Serum hepatic fibrosis indexes
Hepatic histopathologic examination | Change from Baseline at week 24
  Status of the liver
IgG | Change from Baseline at week 24
  Change of humoral immunity
IgA | Change from Baseline at week 24
  Change of humoral immunity
IgM | Change from Baseline at week 24
  Change of humoral immunity
IgE | Change from Baseline at week 24
  Change of humoral immunity
C3 | Change from Baseline at week 24
  Change of humoral immunity
C4 | Change from Baseline at week 24
  Change of humoral immunity
CD3 | Change from Baseline at week 24
  Change of cellular immunity
CD4 | Change from Baseline at week 24
  Change of cellular immunity
CD8 | Change from Baseline at week 24
  Change of cellular immunity
CD19 | Change from Baseline at week 24
  Change of cellular immunity
CD16+56 | Change from Baseline at week 24
  Change of cellular immunity

SECONDARY OUTCOMES:
ALB | Change from Baseline at week 24
  Change of Liver function
ALT | Change from Baseline at week 24
  Change of Liver function
AST | Change from Baseline at week 24
  Change of Liver function
TBIL | Change from Baseline at week 24
  Change of Liver function
DBIL | Change from Baseline at week 24
  Change of Liver function
HBV-DNA | Change from Baseline at week 24
  Status of HBV infection
Change of ultrasound examination of liver | Change from Baseline at week 24
  Status of the liver

CONTACTS AND LOCATIONS:
Overall Officials: YINGAN JIANG, Principal Investigator — Renmin Hospital of Wuhan University
Locations (1):
- Renmin Hospital of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Yes
After approval from the steering committee and the Human Genetic Resources Administration of China, this trial data can be shared with qualifying researchers who submit a proposal with a valuable research question. A contract should besigned.